CLINICAL TRIAL: NCT01296009
Title: Effect of Traditional Chinese Medicine (TCM) on Embryo Implantation in In-vitro Fertilization (IVF) Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Effect of Traditional Chinese medicine (TCM) on embryo implantation in in-vitro fertilization (IVF) patients, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZYF-861234
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2010-11

CONDITIONS: In Vitro Fertilization and Embryo Transfer
Keywords: embryonic implantation; endometrial receptivity; traditional Chinese medicines; in vitro fertilization-embryo transfer; pregnant rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- traditional Chinese medicine (Experimental): The pregnancy rate in traditional Chinese medicine group is higher than the control group
  Interventions: Drug: Traditional Chinese medicine(Zhuyun Recipe)

INTERVENTIONS:
Drug: Traditional Chinese medicine(Zhuyun Recipe) — The patients undergoing IVF-ET take orally traditional Chinese medicine(Zhuyun Recipe) for ten days.

SUMMARY:
To investigate the impact of traditional Chinese medicines (TCM) on embryonic implantation in the patients who have underwent in vitro fertilization and embryo transfer, the investigators compare the pregnancy rate in traditional Chinese medicine group and control group. The hypothesis is that pregnancy rate in traditional Chinese medicine group is higher than the control group.

DETAILED DESCRIPTION:
To demonstrate the impact of traditional Chinese medicine (TCM) on embryo implantation, the investigators perform a prospective randomized study on patients who have underwent in vitro fertilization and embryo transfer (IVF-ET) in the Reproductive Medical Center of the Remin Hospital Wuhan University in the next six months. These patients were randomly divided into two groups, one group was given traditional Chinese medicine, that is, ten days oral administration of Zhuyun recipe from the day after HCG injection. The second group without any treatment, and then the pregnancy rate were observed. Frozen embryo transfer for patients do the same treatment, measured indices were also the same in both groups. Our hypothesis is that Zhuyun recipe is beneficial for embryo implantation in IVF-ET patients, it can be found that pregnancy rate in traditional Chinese medicine group is higher than the control group.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-35 years old
2. undergo IVF/ICSI-ET treatment
3. undergo fresh/ frozen embryos transplantation

Exclusion Criteria:

1. the numbers of embryos transplantation were more than one
2. serum estradiol level > 5000 pg/ml and progesterone level > 9. 54 nmol/L on the day of HCG administration

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | Six months
  12 days after embryo transplantation, the investigators measured blood hCG level in the patients and its level > 10IU/L as a biochemical pregnancy, 4 weeks after transplantation, gestational sac and the beating heart were found as clinical pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Yang, Ph.D, Study Chair — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China